CLINICAL TRIAL: NCT04654715
Title: Surgical and Functional Outcomes of Rectourethral Fistulas Surgery With Gracilis Flap Interposition After Localized Prostatic Cancer Treatment.
Acronym: GRA-FUR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0673
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Rectourethral Fistula
Keywords: rectourethral fistula; Gracilis flap; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Localized prostate cancer treatment induced rectourethral fistula: Every patient over 18 years old operated for closure of a rectourethral fistula with gracilis flap interposition after localized prostatic cancer treatment (Radiotherapy, surgery, cryotherapy and HIFU).
  Interventions: Procedure: Gracilis flap interposition for rectouretral fistula management

INTERVENTIONS:
Procedure: Gracilis flap interposition for rectouretral fistula management — Gracilis flap interposition is a surgery for rectouretral fistula

SUMMARY:
Prostate cancer is the first cancer amongst men with more than 50000 cases per year in France. Surgical, radiation, frost, or ultrasound induced rectourethral fistula is a rare complication (<1%) of localized prostatic cancer treatment but hard to manage. Different types of treatment exist: conservatory, trans-sphinteric (York-Masson), transanal, perineal, with or without muscle flap interposition. Gracilis flap interposition for rectourethral fistula management is a promising technique but few cases are described and functional results are scarce.

The aim of this study is to present surgical and functional outcomes of rectourethral fistulas surgery with gracilis flap interposition after treatment of localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male over 18 years old
* Treated for a localized prostatic cancer (Prostatectomy, cryotherapy, HIFU, radiotherapy)
* Affected with a treatment induced Rectourethral fistula

Exclusion Criteria:

* Rectourethral fistula caused by other pelvic diseases (gynecological or digestif cancer, inflammatory bowel disease, other urogenital issues)
* Rectourethral fistula treated by cysto-prostatectomy with urinary tract derivation
* Patient under guardianship
* Non comprehension of written or spoken French

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients over 18 that have been treated for a localized prostatic cancer and who were affected with a treatment-induced rectourethral fistula
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Urinary continence | 3 months after surgery
  Urinary Symptom Profile form (from 0 to 39), a higher score indicating a worse outcome.
Fecal continence | 3 months after surgery
  St. Marks form (from 0 to 26), a higher score indicating a worse outcome.
Lower extremity functional | 3 months after surgery
  No validated form exist for surgical consequences after gracilis retrieval. The form used in this study is specific (Difficulty scale for walking, kneeling, crossing the legs ; limitation of movements since the operation (yes/no and which one) (From 0 to 20), a higher score indicating a worse outcome.
Surgical scarring | 3 months after surgery
  The Patient and Observer Scar Assessment Scale (From 7 to 70), a higher score indicating a worse outcome.
Global satisfaction of the surgery | 3 months after surgery
  Patients will give a number to measure their global satisfaction of the surgery (From 1 to 10), a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France